CLINICAL TRIAL: NCT02811614
Title: Minimally-invasive Surgery Versus Craniotomy in Patients With Supratentorial Hypertensive Intracerebral Hemorrhage: A Multi-center Randomized Controlled Trial
Brief Title: Minimally-invasive Surgery Versus Craniotomy in Patients With Supratentorial Hypertensive Intracerebral Hemorrhage
Acronym: MISICH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Jingzhou Central Hospital (Other); Wuhan No.1 Hospital (Other); Yichang Central People's Hospital (Other); Second Hospital of Jilin University (Other); The First Affiliated Hospital of Nanchang University (Other); Second Affiliated Hospital of Nanchang University (Other); Tang-Du Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Jiangmen Central Hospital (Other); Jilin Province People's Hospital (Unknown); Siping Central People's Hospital (Other); Minzu Hospital of Guangxi Zhuang Autonomous Region (Unknown); Taihe Hospital (Other)
Responsible Party: Principal Investigator, Xiaolei Chen, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Chinese PLA General Hospital
Record Dates: First submitted 2016-06-20; First posted 2016-06-23 (Estimated); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Intracranial Hemorrhage, Hypertensive
Keywords: intracerebral hemorrhage,hypertensive; minimally invasive surgery; neuroendoscopic surgery; stereotactic aspiration
MeSH Terms: conditions — Intracranial Hemorrhage, Hypertensive | interventions — Craniotomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Experimental 1: Endoscopic Evacuation (Experimental): Endoscopic hematoma evacuation with the help of a self-developed working channel.
  Interventions: Procedure: Endoscopic Evacuation
- Experimental 2: Stereotactic Aspiration (Experimental): Place a catheter into the main body of the hematoma and aspirate blood.
  Interventions: Procedure: Stereotactic Aspiration
- Active Comparator: Craniotomy (Active Comparator): Craniotomy with a big bone flap to for hematoma evacuation.
  Interventions: Procedure: Craniotomy

INTERVENTIONS:
Procedure: Endoscopic Evacuation — Endoscopic surgery for treatment of supratentorial hypertensive intracerebral hemorrhage.
  Other Names: neuroendoscopic surgery
  Arms: Experimental 1: Endoscopic Evacuation
Procedure: Stereotactic Aspiration — Using image guidance to aspirate hematoma.
  Other Names: Hematoma Stereotactic Aspiration
  Arms: Experimental 2: Stereotactic Aspiration
Procedure: Craniotomy — Craniotomy with a big bone flap to evacuate intracerebral hematoma.
  Other Names: Craniotomy evacuation of hematoma
  Arms: Active Comparator: Craniotomy

SUMMARY:
The effectiveness of craniotomy in the treatment of intracerebral hemorrhage remains controversial. Two main types of minimally invasive surgery, endoscopic evacuation and stereotactic aspiration, have been attempted for hematoma removal and show some advantages. However, prospective and controlled studies are still lacking. This is a multi-center randomized controlled trial designed to determine whether minimally invasive hematoma evacuation with endoscopic or stereotactic aspiration will improve the outcome in patients with hypertensive intracerebral hemorrhage compared with small-boneflap craniotomy. Patients will be randomly assigned to endoscopy group, stereotactic aspiration group or small-boneflap craniotomy group in a 1:1:1 ratio.

DETAILED DESCRIPTION:
Hypertensive intracerebral hemorrhage (HICH) is the most common hemorrhagic stroke. The morbidity and mortality exceed 60% and only 12% patients could live independently. The choice of surgical or conservative treatment for patients with HICH is controversial.

Some minimally invasive neurosurgeries have been applied to hematoma evacuation and may improve prognosis to some extent. In endoscopic evacuation, a small burr hole is created and hematoma is removed through suction and irrigation under neuroendoscope. Endoscopic surgical evacuation promise to maximize hematoma evacuation while minimizing damage to normal tissue. Stereotactic aspiration uses image guidance to place a catheter into the main body of the hematoma and aspirate blood. It is estimated that 720 patients (240 patients in each treatment group) would provide 90% power and a type I error probability of .05 to detect an effect size of 13% with a 10% dropout rate taken into consideration. Patients will receive endoscopic evacuation, stereotactic aspiration or craniotomy according to the results of randomization. Patients will be followed up at 7 days, 30 days and 6 months.

Outcomes of different groups of patients will be collected and compared. The study is designed to find a best surgical method for hypertensive intracerebral hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Supratentorial hypertensive intracerebral hemorrhage on CT scan with the hematoma volume ≥25mL
* Adult patients with GCS score ≥5
* Admitted within 24h of ictus

Exclusion Criteria:

* Intracerebral hemorrhage caused by tumor, coagulopathy, aneurysm, or arteriovenous malformation
* Concurrent head injury or history of head injury
* Multiple intracerebral hemorrhage
* Known advanced demential or disability before
* With indications of terminal brain hernia
* Severe concomitant diseases that affect life expectancy
* Patients having taken anti-platelet or anticoagulant drugs for a long time
* With severe intraventricular hemorrhage
* Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 733 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale | 6 months
  The degree of disability or dependence in the daily activities. The scale runs from 0-6, running from perfect health without symptoms to death.

SECONDARY OUTCOMES:
Hematoma Clearance Rate | 24 hours and 3 days
  A ratio assessing extent of hematoma evacuation, ranging from 0 to 100%.
Operation Time | 24 hours
  The time from skin incision to the end of surgery.
Intraoperative Blood Loss | 24 hours
  Volume of blood lost during operation.
Postoperative Glasgow Coma Scale | 7 days
  A neurological scale to record the conscious state of patients at 1 week after surgery.
Rebleeding Rate | 3 days
  The percentage of patients that suffer from rebleeding after surgery. Rebleeding usually occurs within 3 days after surgery.
Days of ICU Stay | 14 days
  The time an ICH patient has to stay in intensive care unit after surgery.
Mortality | 30 days
  The percentage of patients that die within a month after the onset of hypertensive intracerebral hemorrhage.
Intracranial Infection Rate | 7 days
  Percentage of patients that get intracranial infection. The infection should be confirmed by cerebrospinal fluid tests.
Barthel Index | 6 months
  An ordinal scale used to measure performance of patients in activities of daily living. A higher number is associated with a greater likelihood of being able to live at home with a degree of independence following discharge from hospital.
Hospitalization expenses | 6 months
  Total expenses during neurosurgery hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolei Chen, MD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Xu X, Zhang J, Zhang H, Yuan Q, Wang Q, Gan Z, Luo M, Chen X. Efficacy and cost-effectiveness analysis of minimally invasive surgeries for basal ganglia hypertensive intracerebral hemorrhage. J Neurointerv Surg. 2026 Jan 13:jnis-2025-024638. doi: 10.1136/jnis-2025-024638. Online ahead of print. PMID 41529871
- [Derived] Xu X, Zhang H, Zhang J, Luo M, Wang Q, Zhao Y, Gan Z, Xu B, Chen X; MISICH study team. Minimally invasive surgeries for spontaneous hypertensive intracerebral hemorrhage (MISICH): a multicenter randomized controlled trial. BMC Med. 2024 Jun 13;22(1):244. doi: 10.1186/s12916-024-03468-y. PMID 38867192
- [Derived] Xu X, Zheng Y, Chen X, Li F, Zhang H, Ge X. Comparison of endoscopic evacuation, stereotactic aspiration and craniotomy for the treatment of supratentorial hypertensive intracerebral haemorrhage: study protocol for a randomised controlled trial. Trials. 2017 Jun 28;18(1):296. doi: 10.1186/s13063-017-2041-1. PMID 28659171